CLINICAL TRIAL: NCT02293642
Title: Prospective Epidemiology Study to Validate the BOMET-QoL-10 in Patients With Bone Metastasis in Germany
Brief Title: Bone Pain Score Validation Initiative
Acronym: ARIE
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-268
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Bone Metastasis
Keywords: primary cancers of the breast; primary cancers of the kidney; primary cancers of the lung; primary cancers of the prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Translation and validation of the BOMET-QoL-10 questionnaire in Germany and assessment of its validity and responsiveness.

DETAILED DESCRIPTION:
Aim of this study is to translate the questionnaire and to examine the psychometric properties of BOMET-QoL-10 in a German population. Correlations with the EORTC QLQ-C30/BM22 at the time of enrolment and throughout the study aim to verify that the BOMET-QoL-10 is reliable, valid and able to detect stabilization or changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults patients (≥ 18 years)
* Diagnosed cancer of the breast, kidney, lung or prostate
* Bone metastases
* Estimated life expectancy of at least 6 months
* Fluent German speaking, reading and writing
* Informed written consent

Exclusion Criteria:

* Patients without bone metastases
* Participation in another study involving questionnaires
* Patients not able to comply with the assessments specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bone metastases from primary cancers of the breast, kidney, lung or prostate
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
QoL | 6 months
  Validity and responsiveness of the BOMET-QoL-10 questionnaire in reference to EORTC QLQ-C30/BM-22

SECONDARY OUTCOMES:
Impact of characteristics on questionnaire scores | 6 months
  Impact of tumour entity, comorbidity and further parameters on the scores of bone metastasis at baseline
Sensitivity of questionnaire | 6 months
  Sensitivity of BOMET-QoL-10 in patients with / without progression of the disease
Sequence effects of questionnaires | 6 months
  Influence on the order questionnaires are filled out

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Marschner, MD, Principal Investigator — Outpatient Centre for Interdisciplinary Oncology and Haematology, D-Freiburg
Locations (1):
- Multiple Sites All Over Germany, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marschner N, Wilke J, Reschke D, Kaiser F, Schmoor C, Grugel R, Boller E. A brief instrument to measure health-related quality-of-life in patients with bone metastasis: validation of the German version of Bone Metastases Quality-of-Life-10 (BOMET-QoL-10). J Med Econ. 2018 Sep;21(9):920-929. doi: 10.1080/13696998.2018.1484750. Epub 2018 Jun 18. PMID 29874105